CLINICAL TRIAL: NCT06696872
Title: Proprioceptive Neuromuscular Facilitation Versus Core Training for Enhancing Stability and Function in Adolescent With Patellofemoral Pain Syndrome
Brief Title: Enhancing Stability and Function in Adolescent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Amira Hussin Hussin Mohammed, Associated professor, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Patellofemoral Pain Syndrome
Record Dates: First submitted 2024-11-19; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Patellofemoral Pain Syndrome; Adolescents
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core exercises (Experimental): The participants were taught how to contract their deep abdominal muscles to obtain core muscle activation. The patient should be contracting the abdominal muscles, lifting her lower belly up away from pubic bone, while breathing slowly and normally. The patient should not hold her breath
  Interventions: Other: core exercises
- Proprioceptive Neuromuscular Facilitation (Experimental): The hold-relax proprioceptive neuromuscular facilitation stretching protocol consisted of passively moving the dominant leg into a position where the subjects felt mild discomfort and holding that position for 30 seconds. Subjects were then asked to isometrically contract the stretched muscle for 10 seconds; this were followed by muscle relaxation in the same position for 30 seconds, before being stretched to a new point of mild discomfort. The leg were then released
  Interventions: Other: Proprioceptive Neuromuscular Facilitation

INTERVENTIONS:
Other: core exercises — The core muscle strength training program were lasted for 8 weeks and comprised of 3 training sessions per week, with a total of 24 sessions. Each session were lasted for 30 to 45 minutes, starting with a brief warm-up exercise program consisting of low-intensity core strength exercises to prepare the neuromuscular system for the training loads and ending with a cool-down program
  Arms: Core exercises
Other: Proprioceptive Neuromuscular Facilitation — The hold-relax proprioceptive neuromuscular facilitation stretching protocol consisted of passively moving the dominant leg into a position where the subjects felt mild discomfort and holding that position for 30 seconds. Subjects were then asked to isometrically contract the stretched muscle for 10 seconds; this were followed by muscle relaxation in the same posi¬tion for 30 seconds, before being stretched to a new point of mild discomfort. The leg were then released
  Arms: Proprioceptive Neuromuscular Facilitation

SUMMARY:
This study investigated the comparative effects of proprioceptive neuromuscular facilitation (PNF) stretching and core strength exercises on static balance in adolescents with patellofemoral pain syndrome (PFPS).

ELIGIBILITY:
Inclusion Criteria:

* Participants were between 16 and 18 years old.
* Patients had to have experienced anterior knee pain for at least 4 weeks, with the pain being exacerbated by at least two of the following activities: jumping, running, prolonged sitting, stair climbing, kneeling, and squatting (Chevidikunnan et al., 2016).
* Participants could not have undergone any surgical procedures on their lower limbs.
* Pain during the previous week needed to be greater than 30 mm on a 100 mm visual analogue scale (VAS) (Appendix I) (Rathleff et al., 2015).
* A spectrum of BMI was sought, with participants recruited to represent normal BMI percentile categories for both boys and girls. The normal BMI percentile categories for both boys and girls were defined as the 5th percentile to less than the 85th percentile (Appendix II) (King et al., 2012).

Exclusion Criteria:

* Adolescents with cruciate ligament injuries, meniscal injuries, collateral ligament injuries, and tenderness associated with any of these structures, any intra-articular injury, and tenderness over the iliotibial band, patellar tendon, pes anserine tendons, or evidence of joint effusion.

  * Adolescents with referred pain from the hip or lumbar region, or a known case of articular cartilage damage.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS-100 mm) for pain | All adolescents were assessed before and after the 8-week intervention period
Dynamic postural stability test and single leg test using the Biodex Balance System SD | All adolescents were assessed before and after the 8-week intervention period

SECONDARY OUTCOMES:
Self-administered Anterior Knee Pain Scale (AKPS) or Kujala Patellofemoral Score | All adolescents were assessed before and after the 8-week intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Amira H Mohammed, PHD, Principal Investigator — Delta University for Science and Technology
Locations (1):
- Amira Hussin Mohammed, Gamasa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data availability by requesting from the corresponding author and after publication
Time Frame: after 12 months from November 2024